CLINICAL TRIAL: NCT04063059
Title: Women of Color and Family Obesity Management
Brief Title: Black Women's Wellness Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Randall Brown, PI, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BWWP
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Weight, Body; Knowledge, Attitudes, Practice
Keywords: Weight Management; Obesity; African American; Women
MeSH Terms: conditions — Body Weight; Behavior; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Subjects will be randomized to the program intervention which is a female-specific, culturally relevant, self-regulation based in-person group sessions and telephone counseling intervention designed for African American women who are overweight or obese.
  Interventions: Behavioral: PRIDE counseling intervention
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: PRIDE counseling intervention — Step-by-Step program to create positive lifestyle change geared toward wellness and long term healthy living through group sessions and telephone counseling.
  Arms: Intervention

SUMMARY:
The proposed randomized controlled trial will evaluate an educational self-management intervention in 450 African American women and weight management. It will be the first to use a culturally tailored in-person and telephone approach to address all aspects of wellness and social determinants for African American women to achieve optimal long term wellness for both self and family.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American woman, aged 20-59
* BMI 27.5-57.4
* Ability to walk unrestricted for > 3 min
* Caretaker of a child -providing a meal at least 50% of days/week
* Caretaker of at least one child aged 5 -12 years
* Resides in Jackson, Saginaw, Ypsilanti, Lansing, Detroit (All cities in Michigan)
* Speaks English fluently

Exclusion Criteria:

* <12 months postpartum
* Active pregnancy
* Prior or anticipated bariatric surgery
* Non-ambulatory
* History of a severe cardiovascular event (including cerebrovascular accident or myocardial infarction)
* Severe mental illness, neurologic disease and/or cognitive impairment

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Identify as being female
Enrollment: 454 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Weight (lb) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where weight will be collected for all women on the same measurement scale. All measurements will be taken by project staff to ensure data validly.
Weight (lb) | Closing Event (Month 12)
  After 12 months all women will be invited to come to a clinical data collection event "Closing Event" where weight will be collected for all women on the same measurement scale. All measurements will be taken by project staff to ensure data validly.

SECONDARY OUTCOMES:
Height (inches) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where height will be collected for all women on the same stadiometer. All measurements will be taken by project staff to ensure data validly.
Height (inches) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where height will be collected for all women on the same stadiometer. All measurements will be taken by project staff to ensure data validly.
Waist Circumference (inches) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where waist circumference will be collected for all women using the same measuring tape. All measurements will be taken by project staff to ensure data validly.
Waist Circumference (inches) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where waist circumference will be collected for all women using the same measuring tape. All measurements will be taken by project staff to ensure data validly.
Blood Pressure (mmHg) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where blood pressure will be collected for all women using the same electronic blood pressure machine on their non-dominant arm. All measurements will be taken by project staff to ensure data validly.
Blood Pressure (mmHg) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where blood pressure will be collected for all women using the same electronic blood pressure machine on their non-dominant arm. All measurements will be taken by project staff to ensure data validly.
Total Cholesterol (mg/dL) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where total cholesterol will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
Total Cholesterol (mg/dL) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where total cholesterol will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
High Density Lipoprotein Cholesterol (mg/dL) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where High Density Lipoprotein Cholesterol will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
High Density Lipoprotein Cholesterol (mg/dL) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where High Density Lipoprotein Cholesterol will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
Low Density Lipoprotein Cholesterol (mg/dL) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where Low Density Lipoprotein Cholesterol will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
Low Density Lipoprotein Cholesterol (mg/dL) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where Low Density Lipoprotein Cholesterol will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
Triglycerides (mg/dL) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where triglycerides will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
Triglycerides (mg/dL) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where triglycerides will be collected for all women using the same CardioCheck PA Analyzer machine. All measurements will be taken by project staff to ensure data validly.
Hemoglobin A1c | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where Hemoglobin A1c will be collected for all women using the same A1C Now+ machine. All measurements will be taken by project staff to ensure data validly.
Hemoglobin A1c | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where Hemoglobin A1c will be collected for all women using the same A1C Now+ machine. All measurements will be taken by project staff to ensure data validly.
Total Distance Walked (ft) | Kick Off Event (Month 0)
  All women will be invited to come to a clinical data collection event "Kick Off" where women will walk for 6 minutes and total distance will be measured by the same measuring tape. All measurements will be taken by project staff to ensure data validly.
Total Distance Walked (ft) | Closing Event (Month 12)
  All women will be invited to come to a clinical data collection event "Closing Event" where women will walk for 6 minutes and total distance will be measured by the same measuring tape. All measurements will be taken by project staff to ensure data validly.